CLINICAL TRIAL: NCT06346431
Title: Efficacy of Digital Problem Solving Application in Reduction of Anxiety, Depression and Substance Use Disorder Symptoms
Acronym: Efficacy
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: 7 Generation Games (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240301
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Anxiety; Depressive Symptoms; Substance Use Disorders
MeSH Terms: conditions — Anxiety Disorders; Depression; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App Intervention group (Experimental): A project coordinator will meet with the participant to assist in installing the app on device and provide instruction in use. Participants will be able to access support from the app continuously. When in proximity, during service hours to an organization meeting needs identified by the individual, the app will prompt to take action. Data will be collected on symptoms at baseline, three and six months post.
  Interventions: Combination Product: DSPT - Digital Support for Problem-solving Therapy
- Control group (No Intervention): Data will be collected on symptoms at baseline, three and six months post. As individuals have a diagnosis of mental illness they may be receiving "Treatment as usual" for their reservation/ service provider, but no additional services will be provided by the sponsor.

INTERVENTIONS:
Combination Product: DSPT - Digital Support for Problem-solving Therapy — Mobile app breaking major treatment and social needs into subtasks, providing information, prompts and in-app payment to complete those tasks.
  Arms: App Intervention group

SUMMARY:
The focus of this study is the impact of usage of a mobile application to support problem-solving therapy on symptoms of anxiety, depression and substance use.

DETAILED DESCRIPTION:
Tribal communities have a problem. They experience a disproportionate rate of substance use and mental illness. Research shows that customized digital tools designed with the community, integrating local culture and resources are more effective in reducing symptoms of anxiety and depression. However, the cost of design and development renders quality app creation for small markets infeasible. Digital Support for Problem-Solving Therapy in a Tribal Community (DSPT) solves this problem through dramatically reducing software design time by using AI for task analysis and to combine tasks, service programs' geographic coordinates and hours and applying the proprietary 7 Gen Blocks software components to reduce development time. The resulting mobile application will be used by intervention groups on two reservations. At baseline, three months and six months post, both the intervention and randomly assigned control group (total N =100) will complete standardized, validated measures of depression, anxiety and substance use disorder symptoms. All participants will be enrolled members in a federally recognized tribe, over 18 years of age and have a diagnosis of an anxiety, depression or substance use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of anxiety, depression or substance use disorder. Resident on or near Turtle Mountain or Spirit Lake reservation. Enrolled in federally recognized tribe.

Exclusion Criteria:

* Literacy below fourth-grade level. Diagnosis of personality disorder or schizophrenia, or other impaired perception of reality.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder Scale-7 | Six months
  Measure of Anxiety Symptoms
Center for Epidemiological Studies Depression Scale | Six months
  Measure of Depression Symptoms
Drug Abuse Screening Test | Six months
  Screening instrument for abuse of drugs other than alcohol
Michigan Alcohol Screening Test | Six months
  Screening instrument for abuse of alcohol

CONTACTS AND LOCATIONS:
Overall Officials: AnnMaria Demars, Ph.D., Principal Investigator — 7 Generation Games

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] De Mars, A. (2010). Internet usage by Native Americans with Disabilities living on American Indian reservations in the Great Plains. Rural Special Education Quarterly, 29 (2), 34-40.
- [Result] Rousey, A. M. & Longie, E. S. (2001). The tribal college as family support system. American Behavioral Scientist,44 (9), 1492-1504.
- [Result] De Mars, A. & Longie, E. S. (2018). The value of perseverance: Using Dakota culture to teach mathematics. Transmotion, 4 (1), 113-131.